CLINICAL TRIAL: NCT04691349
Title: Chimeric Antigen Receptor T Cells Therapy for r/r Malignant Tumors in Children
Brief Title: CAR-T for r/r Malignant Tumors in Children
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-01
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: CAR-T; Child, Only; Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor T cell (Experimental): Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells. Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner, which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells
  Interventions: Drug: CAR-T

INTERVENTIONS:
Drug: CAR-T — The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region.

SUMMARY:
This study is a clinical study of CAR-T treatment of patients with relapsed/refractory malignant tumors in children. The purpose is to evaluate the safety and effectiveness of chimeric antigen receptor T cells in the treatment of relapsed/refractory malignant tumors in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-18
* Expected survival time ≥ 12weeks
* ECOG 0-2
* At least second-line or above chemotherapy failed
* Liver and kidney function, heart and lung function meet the following requirements:

Creatinine is within the normal range; Left ventricular ejection fraction ≥ 45%; Baseline blood oxygen saturation>91%; Total bilirubin≤1.5×ULN; ALT and AST≤2.5×ULN

* Understand the trial and have signed the informed consent

Exclusion Criteria:

* Those who have graft-versus-host disease (GVHD) or need to use immunosuppressive agents
* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA titer test is not within the normal reference range; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) Antibody positive; CMV DNA test positive; Syphilis test positive
* Severe heart disease
* Systemic diseases judged by the investigator to be unstable: including but not limited to severe liver, kidney or metabolic diseases that require medication
* Within 7 days before screening, there are active infections or uncontrollable infections that require systemic treatment (except for mild urogenital infections and upper respiratory tract infections)
* Those who have received CAR-T therapy or other genetically modified cell therapy before screening
* According to the researcher's judgment, it does not meet the situation of cell preparation
* Situations that other researchers think are not suitable for inclusion

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-01-26 (Estimated); Study Completion 2021-09-26 (Estimated)

PRIMARY OUTCOMES:
ORR3 | Three months after CAR T cell infusion
  3-month objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chilren's Hospital of Soochow University, Suzhou, Jiangsu, China